CLINICAL TRIAL: NCT06389175
Title: Keeping Mind and Body in Sync: Non-invasive Vagus Nerve Stimulation as a Tool to Modulate Stomach-Brain Coupling in Depression
Brief Title: Non-invasive Vagus Nerve Stimulation as a Tool to Modulate Stomach-Brain Coupling in Depression
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Nils B. Kroemer, Prof. Dr. rer. nat., University of Bonn
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BON001; KR 4555/10-1 (Other Grant/Funding Number: Deutsche Forschungsgemeinschaft (DFG))
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Depressive Disorder, Major
Keywords: major depressive disorder; stomach-brain coupling; tVNS
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients suffering from MDD (Experimental): All participants will receive tVNS and sham stimulation in a randomized order.
  Interventions: Device: Transcutaneous non-invasive vagus nerve stimulation (tVNS); Device: Sham stimulation
- Healthy controls (HC) (Experimental): All participants will receive tVNS and sham stimulation in a randomized order.
  Interventions: Device: Transcutaneous non-invasive vagus nerve stimulation (tVNS); Device: Sham stimulation

INTERVENTIONS:
Device: Transcutaneous non-invasive vagus nerve stimulation (tVNS) — Participants receive tVNS during the neuroimaging sessions and the extended stimulation period. To stimulate vagal afferents, the electrode will be placed at the cymba conchae of the right ear using a previously established, conventional stimulation protocol (25 Hz, 30s on/30s off cycle; NEMOS device, Cerbomed, Erlangen, Germany). To improve blinding, the stimulations intensities will be adjusted to correspond to a mild pricking sensation for tVNS and sham.
  The extended stimulation period in the experimental group involves six sessions with at least 1.5h of stimulation (stimulation in the lab or at home with home device using the same stimulation protocol as during the neuroimaging sessions; tVNS R device, tVNS Technologies GmbH, Erlangen, Germany).
Device: Sham stimulation — The control intervention consists of a sham stimulation. In the neuroimaging session the electrode will be placed upside down to stimulate the earlobe, which is not innervated by vagal afferent fibers. To improve blinding, the same stimulation protocol as for the tVNS will be applied (25 Hz, 30s on/30s off cycle; NEMOS device, Cerbomed, Erlangen, Germany) and stimulation intensities will be adjusted to correspond to a mild pricking sensation.
  During the extended stimulation period, the electrode will be placed at the cymba conchae, but only receive a low-intensity stimulation below the perception threshold (0.1mA). To ensure blinding, participants will be instructed that the extended stimulation period will examine the effects of a low- vs. high-intensity tVNS protocol. Each repeated stimulation period will involve six sessions with at least 1.5h of low-intensity stimulation (stimulation in the lab or at home with home device; tVNS R device, tVNS Technologies GmbH, Erlangen, Germany).

SUMMARY:
The overarching goal of the project is to determine whether differences in stomach-brain coupling contribute to key symptoms of major depressive disorder (MDD) and whether transcutaneous non-invasive vagus nerve stimulation (tVNS) may serve as a non-invasive intervention to improve aberrant interoceptive signaling in participants suffering from MDD.

DETAILED DESCRIPTION:
It is planned to conduct a randomized cross-over study including two neuroimaging sessions to assess the effect of acute tVNS (vs. sham) on stomach-brain coupling using concurrent fMRI and EGG. Furthermore, to evaluate potential medium-term effects of repeated applications of tVNS (vs. sham), changes across two weeks in gastric myoelectric frequency and interoception/somatic sensations as well as metabolic and mood states will be evaluated using a combination of lab-based with ecological momentary assessments (EMA).

Consequently, three major hypotheses will be tested:

Hypothesis 1: Participants suffering from MDD show altered stomach-brain coupling compared to matched healthy control participants; inter-individual differences in interoceptive measures/somatic sensations correlate with stomach-brain coupling.

Hypothesis 2: tVNS enhances stomach-brain coupling in a vagal afferent network.

Hypothesis 3: In participants suffering from MDD, tVNS influences interoception/somatic sensations and normalizes gastric myoelectric frequency over an extended stimulation period.

In addition to these main outcomes, tNVS effects on value-based decision-making will be investigated. In detail, participants will be invited to two neuroimaging sessions (T1 and T2) including tVNS or a sham stimulation. At the beginning of each of these sessions, blood will be drawn to determine concentrations of circulating hormones. Afterwards, participants will undergo MRI and complete the following tasks: 1.) Watching an Inscape movie specifically designed to improve imaging at rest. After a 10-minutes baseline scan, tVNS/sham stimulation will start and the Inscape scan is repeated. 2.) Food bidding task to assess neural food cue reactivity as well as bidding behavior and its neural correlates when participants are asked to bid for accessing the presented food. 3.) Foraging task to assess value-based decision-making and its neural correlates with the goal to maximize points in different environments (poor and rich environment). After completing the food bidding and foraging task, the Inscape movie is presented once more to assess tVNS effects after a prolonged stimulation. Throughout all MRI tasks, stomach activity will be assessed by an EGG. Both neuroimaging sessions end with an additional blood draw.

Following the neuroimaging sessions, participants will be invited to two extended stimulation periods (tVNS vs. sham), each lasting approximately two weeks. At the beginning of the extended stimulation periods, participants will be invited to the lab and blood will be drawn (T3). Gastric myoelectric frequency using EGG and value-based decision-making will be assessed at baseline and during stimulation (tVNS or sham). After completing the session, participants are given a tVNS device and are asked to stimulate their vagus nerve for 1.5h at least on four days during the following two weeks. During this time period, participants complete further tasks on value-based decision-making and questionnaires using ecological momentary assessments. In detail, four tasks will cover different aspects of value-based decision making: 1.) Effort allocation task (motivation to work for rewards; completed at T3-T6), 2.) temporal discounting (completed during the whole extended stimulation period), 3.) social discounting (completed during the whole extended stimulation period), and 4.) Influenca (gamified reinforcement learning; completed during the whole extended stimulation period).

After two weeks, participants will again come to the lab and EGG recordings and value-based decision-making tasks will be repeated (T4). Likewise, another blood sample will be collected. The extended stimulation period will then be repeated in the same way for the other stimulation type (tVNS or sham), including both sessions in the lab (T5 and T6). The order of tVNS and sham stimulation is randomized for both neuroimaging sessions as well as the extended stimulation period.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age
* BMI between 18.5 and 30kg/m^2
* Legally valid declaration of consent
* MDD group: current major depressive episode based on DSM V criteria

Exclusion Criteria:

* Current or past diagnosis of brain injury, epilepsy, schizophrenia, bipolar disorder, severe substance use disorder (exception: tobacco), coronary heart disease, stroke
* Following diagnosis within 12 months before start of experiment: obsessive compulsive disorder, somatic symptom disorder, eating disorder
* Contraindications for MRI (e.g. metal implants, claustrophobia) or tVNS (e.g. piercings, sore or diseased skin areas on the outer right ear)
* Pregnant and breastfeeding women are not included
* Unclear ability to give consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Stimulation-induced acute changes in stomach-brain coupling | During MRI scan (up to 120 minutes)
  Stomach-brain coupling will be assessed using phase-locking values (PLV) at baseline and during tVNS/sham stimulation concurrent to electrogastrogram (EGG) measurements in the MRI. PLV will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham) with a focus on core regions of the gastric network (postcentral gyrus, cingulate gyrus, precuneus, occipital cortex, fusiform gyrus, inferior frontal gyrus, inferior and superior parietal lobe, thalamus, and inferior cerebellum) and the vagal afferent pathway (nucleus of the solitary tract (NTS), ventral tegmental area (VTA), substantia nigra, hypothalamus, amygdala, putamen, caudate, nucleus accumbens, hippocampus, insula, ventromedial prefrontal cortex, lateral orbitofrontal cortex, dorsal anterior cingulate cortex). PLV will be correlated with self-reported interoception, somatic symptoms, and depressive symptoms (see below).
Stimulation-induced acute changes in gastric motility | During MRI scan (up to 120 minutes)
  The gastric myoelectric frequency will be assessed during the MRI sessions at baseline and during tVNS and sham stimulation using an EGG. Acute changes in gastric peak frequency will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced mid-term changes in gastric motility | Pre- and post comparison after approx. 2 weeks (beginning and end of extended stimulation period)
  The gastric myoelectric frequency will be assessed at the beginning and end of the extended stimulation periods using an EGG. Data will be collected at baseline and during tVNS and sham stimulation and mid-term changes in gastric peak frequency from the beginning to the end of the extended stimulation periods will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced mid-term changes in self-reported interoception | Pre- and post comparison after approx. 2 weeks (beginning and end of extended stimulation period)
  Interoception is assessed by using the Multidimensional Assessment of Interoceptive Awareness questionnaire, version 2 (MAIA-2). Changes in awareness of bodily sensations will be assessed from the beginning to the end of the extended stimulation period and compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced mid-term changes in somatic symptoms | Pre- and post comparison after approx. 2 weeks (beginning and end of extended stimulation period)
  The Patient Health Questionnaire-15 (PHQ-15) will be used as self-report measurements to assess changes in severity of somatic symptoms from the beginning to the end of the extended stimulation periods. Changes across time will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced mid-term changes in depressive symptoms | Pre- and post comparison after approx. 2 weeks (beginning and end of extended stimulation period)
  The Beck's Depression Inventory (BDI-II) will be used to assess changes in depressive symptoms from the beginning to the end of the extended stimulation periods. Changes across time will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced acute neural changes in food cue reactivity | During MRI scan of a food bidding task (~13 minutes)
  Brain activity (BOLD signal) in response to food stimuli (contrasted with office supplies) and during exerting effort on a grip force device will be analyzed by focusing on brain regions associated with the vagal afferent pathway. Brain activity will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced acute behavioral changes in invigoration | During MRI scan of a food bidding task (~13 minutes)
  Invigoration related to food stimuli (contrasted with office supplies) will be operationalized via the relative effort exerted on a grip force device. Invigoration will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced acute neural changes during foraging | During MRI scan of a foraging task (~25 minutes)
  Brain activity (BOLD signal) during a foraging task will be analyzed by focusing on brain regions associated with the vagal afferent pathway. Brain activity will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced acute behavioral changes in foraging decisions | During MRI scan of a foraging task (~25 minutes)
  Decisions to accept or reject an offered option during a foraging task will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham). Analyses will focus on acceptance rates during different environments (poor and rich environment) for options differing in the effort needed to accept the option and the earned outcome and learning parameters based on trial-to-trial choices.

SECONDARY OUTCOMES:
Stimulation-induced mid-term changes in positive and negative affect | During extended stimulation period (up to approx. 2 weeks)
  Mood will be assessed during the extended stimulation periods via visual analogue ratings (0-100) in ecological momentary assessments. Mood will be surveyed by using items of the Positive and Negative Affect Schedule (PANAS). Changes will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced mid-term changes in self-reported interoception | Pre- and post comparison after approx. 2 weeks (beginning and end of extended stimulation period)
  Participants are asked to indicate their physical sensations on a body silhouette by marking the areas of the body where they perceive activation or deactivation. Interoception is further assessed by using the Visceral Sensitivity Index (VSI). Changes in awareness of bodily sensations will be assessed from the beginning to the end of the extended stimulation period and compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced mid-term changes in motivation | Pre- and post comparison after approx. 2 weeks (beginning and end of extended stimulation period)
  Motivation will be assessed using the effort allocation task at the beginning and the end of the extended stimulation period. Motivation will be operationalized using button press frequency to gain food and monetary rewards. Changes in motivation will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced mid-term changes in physical activity | During extended stimulation period (up to approx. 2 weeks)
  Participants will be asked to wear a smartwatch counting steps and fill out the International Physical Activity Questionnaire (IPAQ) to assess changes in physical activity from the beginning to the end of the extended stimulation periods. Changes will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced mid-term changes in heart rate | During extended stimulation period (up to approx. 2 weeks)
  Participants will be asked to wear a smartwatch to assess changes in heart rate and heart rate variability from the beginning to the end of the extended stimulation periods. Changes will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced acute changes in blood parameters | Before and after stimulation/MRI scan (up to three hours)
  Changes in circulating hormones (e.g., insulin, ghrelin, leptin, glucagon-like peptide-1, cholecystokinin, gastric inhibitory polypeptide) and immune parameters (e.g., C-reactive protein, interleukin 6) will be assessed from blood samples before and after tVNS/sham stimulation during the neuroimaging sessions. Changes will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham). Furthermore, the association of blood parameters with the PLV of the stomach-brain analysis will be evaluated.
Stimulation-induced mid-term changes in blood parameters | Pre- and post comparison after approx. 2 weeks (beginning and end of extended stimulation period)
  Changes in circulating hormones (e.g., insulin, ghrelin, leptin, glucagon-like peptide-1, cholecystokinin, gastric inhibitory polypeptide) and immune parameters (e.g., C-reactive protein, interleukin 6) will be assessed from blood samples at the beginning and end of the extended stimulation period. Changes will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced mid-term changes in composition of microbiome | Pre- and post comparison after approx. 2 weeks (beginning and end of extended stimulation period)
  The bacterial composition of the microbiome as well as the relative frequency of bacterial strains and short-chain fatty acids in the stool will be examined at the beginning and the end of the extended stimulation periods. The first stool sample will be assessed at the beginning of the first stimulation period and a second stool sample will be assessed at the end of the first stimulation period. A this sample will be assessed at the end of the second stimulation period. Changes will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).

OTHER OUTCOMES:
Stimulation-induced mid-term changes in discounting-related decision-making | During extended stimulation period (up to approx. 2 weeks)
  Changes in decision-making during the extended stimulation period will be measured using ecological momentary assessment encompassing temporal and social discounting tasks. Changes will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced mid-term changes in reward learning | During extended stimulation period (up to approx. 2 weeks)
  Changes in reward learning parameters during the extended stimulation period are measured using ecological momentary assessment encompassing a gamified reinforcement learning task (Influenca). Changes will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced mid-term changes in loneliness | During extended stimulation period (up to approx. 2 weeks)
  Changes in self-reported loneliness during the extended stimulation period are measured using ecological momentary assessment. Changes will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).
Stimulation-induced mid-term changes in sleep | During extended stimulation period (up to approx. 2 weeks)
  Participants will be asked to wear a smartwatch to assess changes in sleep (bedtime, rise time, sleep cycles) from the beginning to the end of the extended stimulation periods. Changes will be compared between groups (HC, MDD) and stimulation conditions (tVNS, sham).

CONTACTS AND LOCATIONS:
Overall Officials: Nils B Kroemer, Prof., Principal Investigator — Section of Medical Psychology, Department of Psychiatry & Psychotherapy, Faculty of Medicine, University of Bonn, 53127 Bonn, Germany
Locations (1):
- Section of Medical Psychology, Department of Psychiatry & Psychotherapy, Faculty of Medicine, University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the key results of the study, all anonymized imaging data will be made publicly available (e.g., at openfmri.org)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available after an embargo period of 12 months after completion of the study
Access Criteria: Until the data is publicly available, researchers may contact the lead PI to gain access.
URL: http://neuromadlab.com